CLINICAL TRIAL: NCT02268916
Title: Veterans With Diabetes Mellitus: Improving Physical Activity and Participation
Brief Title: Physical Activity and Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O1190-W
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; physical activity; participation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): OT-led counseling based on home activity pattern
  Interventions: Behavioral: Counseling
- Wait-listed (Placebo Comparator): Usual activity during the study. At the end of the study, will receive OT-led counseling
  Interventions: Behavioral: Usual education

INTERVENTIONS:
Behavioral: Counseling — OT led counseling
  Arms: Intervention
Behavioral: Usual education — At the end of the study, will receive OT-led counseling
  Arms: Wait-listed

SUMMARY:
The purpose of the study is to investigate if the investigators can improve physical activity and social participation level among Veterans with diabetes.

DETAILED DESCRIPTION:
Physical activity is the cornerstone of good diabetes management, and yet effective physical activity intervention is not available. The investigators developed a lifestyle intervention based on individual's home activity patterns. The goal of the study is to test the efficacy of this intervention among Veterans with diabetes in a randomized-controlled trial. In addition to physical activity, the investigators will also assess if the intervention will improve social participation among Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Aged 60 years or older
* Has Type 2 diabetes mellitus
* Able to operate accelerometer
* Competent to consent to the study
* No dementia diagnosis
* Ambulatory with or without assistive device
* English-speaking
* Community living (i.e., not a nursing home resident)
* Not physically active on a regular basis (less than 150 minutes of moderate or vigorous physical activity per week)

Exclusion Criteria:

* Medically unstable
* Hospitalized within the last 6 months
* 2 or more days of complete bed rest in the last month
* hemiplegia or limb amputation
* Self-reported illness or conditions that would impair the cooperation with the study team or the ability to complete the study
* work involved in shift schedule
* current enrollment of a physical activity program
* replacement of hip or knee within the last 6 months.
* Parkinson's disease
* frequent falls

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pearl G. Lee, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Wait-listed
Started | 52 | 52
Completed | 35 | 42
Not Completed | 17 | 10
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Participant did not have diabetes | 1 | 0
Not completed — Did not complete home monitoring activities after baseline visit | 9 | 4

BASELINE CHARACTERISTICS:
Population: One participant was identified to not have diabetes diagnosis after consent, therefore, no baseline data collected on this participant and s/he was not included in further analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait-listed | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 49 | 47 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.83 (5.55) | 71.54 (6.73) | 72.14 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 51 | 50 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 44 | 41 | 85
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 52 | 103

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: Home physical activity changes from baseline to 6-months.Physical activity was measured using a validated survey called CHAMPS, asking the participants to report activities that they participated in a typical week, such as walking, doing house work, dancing, etc.
Time Frame: 6 months
Population: Only participants who completed the home monitoring activities were included in the outcomes analysis.
Measure: Mean (Standard Deviation); unit: KCal/week
Arm/Group | Intervention | Wait-listed
Number analyzed (Participants) | 35 | 42
KCal/week | 401.88 (3909.59) | -263.81 (4414.79)
Statistical Analysis 1: Comparison: Intervention vs Wait-listed; We hypothesized that at the end of 6 months, the intervention group will have increased physical activity as measured by CHAMPS compared to the control group; Test type: Superiority — The study was powered based on a two-sample t-test of the primary outcomes, changes in physical activity or social participant over 6 months. Based on previous literature, in order to detect an effect size of 0.28 with at least 70% power, we aimed to recruit at least 35 participants in each treatment group; p = 0.18, Mixed Models Analysis; The outcome was adjusted for time of visit, visit x intervention group, age, gender, body mass index, insulin, depression, and time-up-and-go score; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-0.18 to 0.97]

2. Primary Outcome: Social Participation
Description: Survey questionnaires of participation change from baseline to 6-months follow up, specifically, satisfaction with participation in social roles, satisfaction with participation in discretionary social activities, and ability to participate in social roles and activities. Each survey has been validated and scored on the T-score metrics. A T-score is a standardized score, and has a "middle" score; it is 50 for T-scores. This middle score is the mean of a large sample that is representative of the US general population. The survey results are T-score metrics in which 50 is the mean score of the general population and 10 is the standard deviation (SD) of that population. The study outcomes are changes in T-scores of each survey from baseline to 6-months follow-up, where positive score means improved outcome, and negative score means worse outcome at 6-months.
Time Frame: 6 months
Population: Only participants with completed surveys were included in the analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention | Wait-listed
Number analyzed (Participants) | 35 | 42
T-score
  Satisfaction social roles | 0.18 (7.47) | 0.63 (8.43)
  Satisfaction discretionary social roles | 0.35 (8.14) | 0.85 (7.29)
  Ability to participate social roles and activities: number analyzed (Participants) | 33 | 42
  Ability to participate social roles and activities | -0.55 (7.50) | -0.36 (7.40)
Statistical Analysis 1: Comparison: Intervention vs Wait-listed; We hypothesized that at the end of 6 months, intervention group will have improved participation as measured by satisfaction with participation in social roles; Test type: Superiority; p = 0.19, Mixed Models Analysis; Slope = -2.20, 95% CI 2-sided [-5.45 to 1.06]
Statistical Analysis 2: Comparison: Intervention vs Wait-listed; We hypothesized that at the end of 6 months, intervention group will have improved participation as measured by satisfaction with participation in discretionary social activities; Test type: Superiority; p = 0.57, Mixed Models Analysis; Slope = -1.02, 95% CI 2-sided [-4.53 to 2.48]
Statistical Analysis 3: Comparison: Intervention vs Wait-listed; We hypothesized that at the end of 6 months, intervention group will have improved participation as measured by the survey on the ability to participate in social roles and activities; Test type: Superiority; p = 0.12, Mixed Models Analysis; Slope = -2.44, 95% CI 2-sided [-5.52 to 0.63]

3. Other Pre Specified Outcome: Physical Function
Description: Six month changes in timed up and go test, where the participant get up from sitting in a chair, walk meters, turn around, and walk back to sit down. Positive changes means worse outcome for timed up and go (seconds).
Time Frame: 6 months
Population: Only participants who completed the 6-months physical function assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention | Wait-listed
Number analyzed (Participants) | 32 | 38
seconds | 0.01 (1.68) | -0.25 (2.69)
Statistical Analysis 1: Comparison: Intervention vs Wait-listed; We hypothesized that at 6-month follow-up, the intervention group will have better performance than the control group in timed up and go test; Test type: Superiority; p < 0.05, Mixed Models Analysis; Slope = -1.99, 95% CI 2-sided [-3.97 to -0.02]

4. Other Pre Specified Outcome: Physical Function
Description: Six month changes in gait speed, which is the comfortable gait peed in 10 meter walking. Positive changes means better outcomes for gait speed (meters per second).
Time Frame: 6 months
Population: Only participants who completed the 6-months physical function assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: meter per second
Arm/Group | Intervention | Wait-listed
Number analyzed (Participants) | 32 | 38
meter per second | 0.01 (0.14) | 0.00 (0.11)
Statistical Analysis 1: Comparison: Intervention vs Wait-listed; We hypothesized that at 6-month follow-up, the intervention group will have better performance than the control group in gait speed; Test type: Superiority; p = 0.02, Mixed Models Analysis; Slope = 0.11, 95% CI 2-sided [0.02 to 0.20]

5. Other Pre Specified Outcome: Physical Function
Description: Six month changes in six-minute walk test, which measures the distance a participant walked at usual pace for six minutes. Positive changes means better outcomes for six-minute walk (meters).
Time Frame: 6 months
Population: Only participants who completed the 6-months physical function assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention | Wait-listed
Number analyzed (Participants) | 32 | 36
meters | 4.23 (45.97) | 5.19 (35.73)
Statistical Analysis 1: Comparison: Intervention vs Wait-listed; We hypothesized that at 6-month follow-up, the intervention group will have better performance than the control group in six-minute walk test; Test type: Superiority; p = 0.02, Mixed Models Analysis; Slope = 40.04, 95% CI 2-sided [7.90 to 72.17]

ADVERSE EVENTS:
Time Frame: For each participant, the adverse event data were collected from the beginning of the enrollment until the last follow up visit, up to 6-months final follow up visit, or when the participant withdrew from the study. For the wait-list group, the participants may complete the OT-intervention up to one month after the 6-months follow-up visit, thus the total follow up period may be 7 months.
Groups:
- Wait-listed Without OT-Led Counseling: Usual activity during the study. At the end of the study, will receive OT-led counseling
  Usual education
- Wait-listed With OT-Led Counseling: Usual activity during the study. At the end of the study, will receive OT-led counseling
  Counseling: At the end of the study, will receive OT-led counseling
Arm/Group | Intervention | Wait-listed Without OT-Led Counseling | Wait-listed With OT-Led Counseling
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 2/52 | 0/52 | 1/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=52) | Wait-listed Without OT-Led Counseling (N=52) | Wait-listed With OT-Led Counseling (N=52)
Minor , possibly study related adverse events (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Muscle sprain, knee pain
Minor, possibly study related adverse events (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — A fall under unclear circumstances and did not need to seek medical care
Minor, possibly related to the study (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — toe nail bleed may be related to walking

LIMITATIONS AND CAVEATS:
The study participants are predominantly male and are all veterans, so the results would be difficult to be generalized to female and non-veterans. Physical activity is measured by a survey, which may have recall bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT02268916/Prot_SAP_000.pdf